CLINICAL TRIAL: NCT00004032
Title: Intraperitoneal (IP) Autologous Therapeutic Tumor Vaccine AUT-OV-ALVAC-h.B7.1 Plus IP rIFN-gamma for Patients With Ovarian Cancer. A Pilot Study
Brief Title: Tumor Vaccine and Interferon Gamma in Treating Patients With Refractory Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02255; MDA-ID-96253; U01CA062461 (NIH); CDR0000065850 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-12-10; First posted 2003-08-25 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Ovarian Epithelial Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Interferon-gamma; interferon gamma-1b

ARMS (1):
- Treatment (ALVAC-hB7.1, recombinant interferon gamma) (Experimental): Patients receive ALVAC-hB7.1 infected tumor cells intraperitoneally (IP) on days 4, 11, and 18. Patients also receive interferon gamma IP on days 8, 10, 15, and 17. In the absence of disease progression, up to 6 courses of therapy may be given. If insufficient tumor cells are available to continue treatment with tumor cell derived vaccine, interferon gamma may be given alone.
  Interventions: Biological: ALVAC-hB7.1; Biological: recombinant interferon gamma; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: ALVAC-hB7.1 — Given IP
Biological: recombinant interferon gamma — Given IP
  Other Names: Actimmune; gamma interferon; IFN-G
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase I trial to study the effectiveness of a tumor cell vaccine and interferon gamma in patients with refractory epithelial ovarian cancer. Vaccines made from a person's cancer cells may make the body build an immune response to and kill their tumor cells. Combining vaccine therapy with interferon gamma may be a more effective treatment for epithelial ovarian cancer

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine whether intraperitoneal (IP) injections of epithelial ovarian carcinoma cells infected with ALVAC-hB7.1 and IP interferon gamma have acceptable toxicity and produce any clinical responses in patients with refractory ovarian epithelial cancer.

OUTLINE: This is a dose-escalation study of ALVAC-hB7.1 infected tumor cells.

Patients receive ALVAC-hB7.1 infected tumor cells intraperitoneally (IP) on days 4, 11, and 18. Patients also receive interferon gamma IP on days 8, 10, 15, and 17. In the absence of disease progression, up to 6 courses of therapy may be given. If insufficient tumor cells are available to continue treatment with tumor cell derived vaccine, interferon gamma may be given alone. Cohorts of 3 to 6 patients receive escalating doses of ALVAC-hB7.1 infected tumor cells until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 6 months until disease progression.

PROJECTED ACCRUAL: A total of 12 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ovarian epithelial carcinoma
* Previously treated with an adequate course of platinum based chemotherapy
* Evidence of intraabdominal disease
* No significant adhesions
* Performance status - Zubrod 0-2
* Lymphocyte count at least 500/mm^3
* Bilirubin no greater than 1.5 mg/dL
* SGOT less than 2.5 times upper limit of normal
* Creatinine no greater than 1.5 mg/dL
* No major disorder of the cardiovascular system
* No major disorder of the pulmonary system
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Successful placement of peritoneal catheter
* No overt autoimmune disease
* No concurrent chronic steroid therapy
* No prior radiotherapy
* Prior surgery allowed
* Recovered from prior therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 1997-10; Primary Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Autologous tumor cell cytotoxicity lymphocyte (CTL) | Up to 7 years
Cytokine production (IFN gamma, IL-10, IL-2) by RT-PCR | Up to 7 years
Toxicity as assessed by NCI Common Terminology Criteria (CTC) | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Freedman, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States